CLINICAL TRIAL: NCT05506631
Title: Cost of Inpatient Care for Women Undergoing Outpatient vs. Inpatient Transcervical Balloon Cervical Ripening for Induction of Labor at Term
Brief Title: Foley Balloon Study for Cervical Ripening - Cost Comparison Between Outpatient and Inpatient Cervical Ripening
Acronym: Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Joanne Quinones, MD, Vice Chair Research, Dept OBGYN, Lehigh Valley Health Network, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000949
Record Dates: First submitted 2021-12-08; First posted 2022-08-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Outcome
Keywords: cervical Ripening; Labor, induced; Term Birth

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient cervical ripening (Experimental): Placement of transcervical Foley balloon for cervical ripening in outpatient setting
  Interventions: Procedure: Outpatient Foley balloon placement
- Inpatient cervical ripening (Active Comparator): Placement of transcervical Foley balloon for cervical ripening in inpatient setting
  Interventions: Procedure: Inpatient Foley Balloon placement

INTERVENTIONS:
Procedure: Outpatient Foley balloon placement — Cervical ripening with balloon placement in the outpatient setting
  Arms: Outpatient cervical ripening
Procedure: Inpatient Foley Balloon placement — Cervical ripening with balloon placement in the inpatient setting
  Arms: Inpatient cervical ripening

SUMMARY:
The objective of this study is to determine the impact of outpatient cervical ripening with transcervical balloon placement for induction of labor at term on the length and cost of inpatient hospitalization when compared to inpatient cervical ripening.

DETAILED DESCRIPTION:
The objective of the study is to determine the impact of outpatient cervical ripening with transcervical balloon placement for induction of labor at term on the length and cost of inpatient hospitalization when compared to inpatient cervical ripening.

Specific Aims

In conducting this study, the investigators will accomplish the following specific aim:

To compare the length of inpatient care for women undergoing cervical ripening with a transcervical Foley placed in the outpatient vs. inpatient setting prior to induction of labor.

* Primary outcomes of interest
* The length of time (measured in minutes) spent on the inpatient unit (L&D) from admission for cervical ripening and/or labor induction until delivery.

Outpatient arm:

Time for the participants in the outpatient group will be measured from the time the participant is admitted to the hospital for induction of labor until she delivers.

Inpatient arm:

Time for the participant in the inpatient group will be measured from the time the participant is admitted to the hospital for cervical ripening with balloon placement and induction until she delivers.

Time from admission to L&D until delivery = total INPATIENT until delivery (hours)

• Cost Analysis

Cost/charges will be calculated for the time spent in the outpatient and inpatient unit for both randomization groups.

Cost will be based on information obtained from Enterprise Analytics charges for the time each participant spends in outpatient care, inpatient care, hospitalized from admission to the L&D unit to delivery.

The investigators will report on the delta/difference in average costs of outpatient and inpatient care between the outpatient and inpatient arms of the study.

Information will be obtained from the finance department at LVHN.

* Secondary outcomes of interest to be compared by randomization groups include:
* maternal outcomes
* mode of delivery, chorioamnionitis, endometritis, placental abruption, urinary tract infection, preeclampsia, wound infection, venous thromboembolism, maternal treatment with postpartum antibiotics
* neonatal outcomes
* neonatal birthweight, Apgar scores, admission to the neonatal intensive care unit (ICU), neonatal ICU length of stay, neonatal hypoglycemia, neonatal sepsis, neonatal seizures, meconium aspiration, intubation for respiratory support, neonatal length of stay (total), umbilical cord gas pH, neonatal death or stillbirth
* dosing of narcotic medications before regional anesthesia
* total oxytocin infusion dosing
* total length of stay for mothers and neonates

ELIGIBILITY:
Inclusion Criteria

* Pregnant women at ≥39 weeks gestation by reliable dating criteria as determined by the American College of Obstetricians and Gynecologists
* Scheduled induction of labor with indication and timing supported by Lehigh Valley Health Network -Labor and Delivery Units (Cedar Crest & Muhlenberg)
* Singleton gestation
* Cephalic presentation
* Amniotic fluid index normal
* Formal prenatal ultrasound during the pregnancy documenting the absence of placenta previa
* Bishop score <6 and cervical dilation <3cm at the time of decision to induce labor
* The woman is able to give appropriate consent and has undergone an informed consent process.
* Maternal age ≥ 18 years old at the time of consent
* English speaking

Exclusion Criteria

* Undergoing outpatient antenatal testing for any medical or obstetric condition
* Need for inpatient observation or continuous fetal monitoring during their cervical ripening
* New diagnosis requiring immediate hospitalization for monitoring (such as new onset hypertensive disease of pregnancy)
* Vaginal bleeding
* Active labor
* Premature rupture of membranes
* Uterine tachysystole (>5 contractions in 10 minutes)
* Non-reassuring fetal heart tracing before Foley placement
* Intrauterine fetal demise diagnosed after enrollment and before placement of balloon
* Contraindication to vaginal delivery, relative or absolute (i.e. transfundal uterine surgery)
* Abnormal placentation including a low lying placenta
* Prior cesarean delivery
* Known fetal major anomaly
* Human immunodeficiency virus, Hepatitis C, or active herpes infection
* Maternal cardiopulmonary disease requiring cardiac monitoring during labor
* Pregestational diabetes or GDMA2
* Rh isoimmunization
* Non-English speaking
* BMI > 40
* Distance from the hospital over 60 minutes by car, unreliable communication via telephone, or unreliable transportation

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
The length of time (measured in minutes) spent on the inpatient unit from admission from cervical ripening and/or labor induction until delivery. | 12 months
  The length of time (measured in minutes) spent on the inpatient unit (L&D) from admission for cervical ripening and/or labor induction until delivery.
Cost Analysis in dollars Cost/charges will be calculated for the time spent in the outpatient and inpatient unit for both randomization groups. | 12 months
  Cost Analysis in dollars
  Cost/charges will be calculated for the time spent in the outpatient and inpatient unit for both randomization groups.
  Cost will be based on information obtained from Enterprise Analytics charges for the time each woman spends in outpatient care, inpatient care, hospitalized from admission to the L&D unit to delivery.

SECONDARY OUTCOMES:
Delivery | 12 months
  Mode of Delivery
Maternal state | 12 months
  Maternal outcomes
Neonatal State | 12 months
  Neonatal outcomes
Maternal Adverse events | 12 months
  Maternal Adverse events such as chorioamnionitis; endometritis; placental abruption; urinary tract infection; preeclampsia,; wound infection; venous thromboembolism; need for post partum antibiotics
Neonatal adverse events | 12 months
  Neonatal Adverse events such as: hypoglycemia; sepsis; seizures; meconium aspiration; respiratory failure; death
Birthweight | 12 months
  neonatal birthweight in kilograms
ICU Length of stay | 12 months
  neonatal ICU length of stay in days
Total Length of stay | 12 months
  neonatal Inpatient length of stay in days
Cord PH | 12 months
  Umbilical cord gas PH as reported
Narcotic dosing | 12 months
  Maternal dosing of narcotic medications before regional anesthesia
Oxytocin dosing | 12 months
  Oxytocin dose per unit
Maternal length of stay | 12 months
  Maternal inpatient length of stay in days

CONTACTS AND LOCATIONS:
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States